CLINICAL TRIAL: NCT03370588
Title: The Influence of Perioperative Administration of Dexmedetomidine on Inflammation Response and Postoperative Outcomes in Patients Undergoing Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Cytoreductive Surgery; Double Blind Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2017-0372
Record Dates: First submitted 2017-11-21; First posted 2017-12-12 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Investigator prepared the drug and participant and outcomes assessor were blind to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine infusion group (Experimental)
  Interventions: Drug: dexmedetomidine
- normal saline infusion group (Active Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: dexmedetomidine — Group A: dexmedetomidine infusion (0.4㎍/kg/hr) from anesthetic induction until the start of closure of peritoneum. Group B: Saline infusion during same time period.
  Arms: dexmedetomidine infusion group
Drug: Normal saline — Group B: Saline infusion during same time period.
  Arms: normal saline infusion group

SUMMARY:
Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) has been reported to be an effective treatment approach for peritoneal cancer, however, the stress response to HIPEC is major neuroendocrine and cytokine response, which has been considered as the homeostatic defense mechanism. Recently, dexmedetomidine has been suggested to exhibit anti-inflammatory properties. This study was designed to evaluate the effect of perioperative administration of dexmedetomidine on inflammation response and postoperative outcomes in patients undergoing hyperthermic intraperitoneal chemotherapy (HIPEC) cytoreductive surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients between 20 and 70 years old
* obtaining written informed consent from the patients who were undergoing hyperthermic intraperitoneal chemotherapy (HIPEC) cytoreductive surgery
* weights under 90 kg and BMI under 32

Exclusion Criteria:

* emergency operation
* re-operations
* combined surgery over 4 departments.
* cardiac disease (unstable angina, congestive heart failure, valvular heart disease)
* Ventricular conduction abnormality
* prior pacemaker insertion
* uncontrolled hypertension (diastolic blood pressure > 110mmHg)
* bradycardia (HR < 40 Bpm)
* cerebral vascular disease (cerebral hemorrhage, cerebral ischemia)
* hepatic or renal failure
* patients who take antiarrythmic agent
* neurological or psychiatric illnesses
* foreigner and patient who can not read the letter

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
IL-6 level | Up to 12 hours after surgery
  To evaluate the effect of dexmedetomidine on the level of IL-6 in patient undergoing HIPEC, IL-6 level was measured up to 12 hours after surgery.

SECONDARY OUTCOMES:
recurrence rate | up to 1 year after surgery
  To evaluate the effect of dexmedetomidine on the recurrence rate up to 1 year after surgery were collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No